CLINICAL TRIAL: NCT03613636
Title: The Role of Adaptive Immune Responses to Mycoplasma Pneumoniae in Pathogenesis and Diagnosis of Community-acquired Pneumonia (CAP) in Children: an Observational Single-center Study (myCAP Study)
Brief Title: Evaluation of Pathogenesis and Diagnosis of Mycoplasma Pneumoniae Community-acquired Pneumonia (CAP)
Acronym: myCAP
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-00148
Record Dates: First submitted 2018-07-06; First posted 2018-08-03 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Childhood Pneumonia; Mycoplasma Pneumonia; Antibody-secreting Cells; Enzyme-linked Immunospot (ELISpot); Diagnosis
MeSH Terms: conditions — Pneumonia, Mycoplasma; Disease | interventions — Enzyme-Linked Immunospot Assay; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Respiratory samples (pharyngeal swab specimens);
  * Peripheral venous bood (peripheral blood mononuclear cells (PBMCs) and serum).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CAP cohort: * Children of age 3 to 16 years;
  * In- and outpatients;
  * Clinically diagnosed community-acquired pneumonia (CAP).
  Interventions: Diagnostic Test: Enzyme-linked immunospot (ELISpot) assay [Blood]
- Healthy control cohort: * Healthy asymptomatic children of age 3 to 16 years;
  * undergoing an elective surgical procedure.
  Interventions: Diagnostic Test: Enzyme-linked immunospot (ELISpot) assay [Blood]
- Family control cohort: - Family members of index CAP patients.
  Interventions: Diagnostic Test: Enzyme-linked immunospot (ELISpot) assay [Blood]

INTERVENTIONS:
Diagnostic Test: Enzyme-linked immunospot (ELISpot) assay [Blood] — The ASC ELISpot will be developed based on the improved methods recently described [Nat Protoc 2013;8:1073-87]. This protocol allows rapid (6-8 h) detection of specific ASCs in small volumes (1-2 ml) of blood. M. pneumoniae protein P1 (50 μl/ml) will be used as antigen. The optimal concentration of coating antigen will be assessed in advance in two-fold serial dilutions for clear spot definition. The M. pneumoniae-specific T cell ELISpot will be developed based on methods recently described [Nat Protoc 2009;4:461-9].
  Other Names: Polymerase chain reaction (PCR) [Pharyngeal swab specimens]; Enzyme-linked immunosorbent assay (ELISA) [Serum]

SUMMARY:
To investigate the Mycoplasma pneumoniae-specific circulating antibody-secreting cell (ASC) response and Mycoplasma pneumoniae-specific interferon (INF)-γ-secreting T cell response, along with polymerase chain reaction (PCR) and serology, in a cohort of children with community-acquired pneumonia (CAP) and controls.

ELIGIBILITY:
Inclusion Criteria:

CAP cohort:

* Children of age 3 to 18 years;
* In- and outpatients;
* Clinically diagnosed community-acquired pneumonia (CAP);

Healthy control cohort:

- Healthy asymptomatic children of age 3 to 18 years undergoing an elective surgical procedure;

Family control cohort:

- Family members of index CAP patients.

Exclusion Criteria:

* Hospital-acquired pneumonia;
* Immunodeficiencies;
* Chronic lung disorders.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: CAP cohort:
  There will be a consecutive ongoing recruitment through the project leader or instructed physicians of the department of infectious diseases and emergency in daily clinical practice.
  Healthy control cohort:
  The project leader will be informed by the local surgeons about a planned elective surgical procedure, unrelated to respiratory tract disease, and will include children during the pre-operation discussion. Samples will be collected by the anaesthesist prior to the start of the surgical procedure, while the child is under general anaesthesia and has an intravenous line. In a subgroup of such children undergoing planned adenotomy, the removed adenoids will be collected after surgery.
  Family control cohort:
  Family members will be included simultaneously with the index CAP patients.
Sampling Method: Probability Sample
Enrollment: 490 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Change in numbers of M. pneumoniae-specific ASCs and M. pneumoniae-specific INF-γ-secreting T cells in blood from inclusion (day 0) to 1-month follow-up (day 28) | At day 0 (inclusion, disease presentation) and at day 28 (follow-up, disease resolution)
  Enzyme-linked immunospot (ELISpot) assay and flow cytometry

SECONDARY OUTCOMES:
Change in M. pneumoniae DNA levels in respiratory samples from inclusion (day 0) to 1-month follow-up (day 28) | At day 0 (inclusion, disease presentation) and at day 28 (follow-up, disease resolution)
  PCR
Change in total and M. pneumoniae-specific antibody levels (immunoglobulin (Ig)G, IgM, IgA) from inclusion (day 0) to 1-month follow-up (day 28) | At day 0 (inclusion, disease presentation) and at day 28 (follow-up, disease resolution)
  Enzyme-linked immunosorbent assay (ELISA)
Outcome of community-acquired pneumonia (CAP) assessed by clinical assessment of body temperature (°C) and respiratory rate (per minute) at 1-month follow-up (day 28) | At day 28 (follow-up)
  Clinical assessment of body temperature (°C) and respiratory rate (per minute), with worse outcome defined as body temperature more than 38.5°C and respiratory rate according to age more than 40/min for 3 years, more than 34/min for 4-5 years, more than 30/min for 6-12 years, and more than 16/min for 13-18 years.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick M. Meyer Sauteur, MD, Principal Investigator — University Children's Hospital, Zurich

IPD SHARING:
Plan to Share IPD: Undecided
Not yet defined.